CLINICAL TRIAL: NCT00616356
Title: Characterization of T Cell Responses Following Yellow Fever Virus Vaccination in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Charles Rice, Professor, Rockefeller University
Other Study IDs: RUH IRB # CRI-0618
Record Dates: First submitted 2008-01-23; First posted 2008-02-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Yellow Fever
Keywords: Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators at Rockefeller University are doing this research to study how the immune system responds to viruses and other infectious agents by using the yellow fever 17D vaccine as a model. The YFV-17D vaccine is one of the safest and most effective vaccines known and has been used to vaccinate humans against yellow fever virus (YFV) infection since the 1930s. By studying how the human immune system responds to the YFV vaccine we hope to learn more about the normal functioning of the immune system so that it might be possible to design new, more effective types of vaccines to prevent important infectious diseases.

The reason for doing this research is:

Currently there is very little information about which factors determine the effectiveness of the initial (primary) immune response to a foreign substance (antigen), such as a virus, that person may be exposed to. There is also very little known about what determines how effectively and for how long a person's immune system can react to the same antigen to prevent another infection. Studies in animals have given us important information about how the immune systems of other animals behave upon initial or repeated exposure to antigens,but these topics have not been studied in detail in humans.

The following hypotheses will be tested:

* The magnitude of the initial expansion of T lymphocytes (the "clonal burst") specific for the infecting virus determines the level at which memory T cell responses are generated against the specific viral antigen and the duration of the memory T cell response generated in the body.
* The majority of CD8 T cells generated after immunization are yellow fever specific and not "bystander activation" of non-specific cells.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Age 18-45 years.
3. Agrees not to take any vaccines within 30 days before or 30 days after YFV vaccination.

Exclusion Criteria:

1. Previously vaccinated with yellow fever vaccine.
2. A history of a medical condition resulting in impaired immunity.
3. Use of immunosuppressive medications.
4. Thymus gland dysfunction.
5. Recipient of a blood product or immune globulin product within 42 days of the screening visit or 30 days after the YFV vaccination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Rockefeller University Personnel
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Rice, PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States